CLINICAL TRIAL: NCT01733069
Title: Clinical Evaluation of the APTIMA® COMBO 2®Assay Using the PANTHER™ System
Brief Title: Clinical Evaluation of the APTIMA® COMBO 2® Assay Using the PANTHER™ System
Status: Completed | Type: Observational
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: AC2PS-US11-001; ACTPS-US10-001 (Other: Gen-Probe)
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-11

CONDITIONS: Chlamydia Trachomatis; Neisseria Gonorrhoeae Infection
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 4 specimens will be collected from each female subject in the following order: 1 first-catch urine specimen, 1 vaginal swab specimen (patient or clinician-collected), 1 cervical specimen (using a broomlike collection device or a brush/spatula combination), and 1 endocervical swab specimen. An additional cervical specimen may be collected from female subjects for other clinical trial purposes or research studies. Up to 2 specimens will be collected from each male subject in the following order: 1 urethral swab specimen and 1 first-catch urine specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment
  Interventions: Device: APTIMA COMBO 2 Assay (AC2 Assay)

INTERVENTIONS:
Device: APTIMA COMBO 2 Assay (AC2 Assay) — APTIMA COMBO 2 Assay (AC2 Assay

SUMMARY:
The objectives of this study are to establish the performance characteristics of the AC2 (APTIMA Combo 2) Assay on the PANTHER System for the sample types cleared for use on the TIGRIS and DTS (Direct Tube Sampling) Systems and to demonstrate the repeatability and reproducibility of the AC2 Assay on the PANTHER System.

DETAILED DESCRIPTION:
The results of this protocol AC2PS-US11-001 (NCT01733069) are based on samples collected from protocol ACTPS-US10-001(NCT01358799).

The registration for NCT01358799 was withdrawn because the samples were not tested under protocol ACTPS-US10-001, instead they were tested under the protocol registered here AC2PS-US11-001 (NCT01733069).

ELIGIBILITY:
Inclusion Criteria:

•The subject is at least 14 years of age at the time of informed consent and is sexually active

* The subject reports symptoms consistent with a suspected STD (sexually transmitted disease) such as abnormal discharge, genital itching, pain/discomfort during sexual intercourse or urination, and/or lower abdominal discomfort.
* If the subject is asymptomatic, the subject is known to be partners with, or a contact of, a person with a confirmed or suspected STD(s), is undergoing screening evaluation for a possible STD(s), and/or is scheduled for a routine exam that may include a pelvic exam
* The subject and/or legally authorized representative is willing to undergo the informed consent process prior to study participation (a minor will need the documented consent of his/her parent or legal guardian, unless the site has an IRB (institutional review board) approved waiver for parental consent for minors)

Exclusion Criteria:

•A potential subject will be ineligible for clinical trial enrollment if the subject, clinician, or medical record reports any of the following:

* The subject took antibiotic medications within the last 21 days
* The subject is underage (as defined by the IRB (institutional review board) or state law), without the documented consent of her/his parent or legal guardian (exception: sites that have an IRBapproved waiver for parental consent for minors)
* The subject is determined by the investigator to be medically unsuitable for participation in this study (eg, medical history of concurrent illness that could result in an unacceptable risk to the subject) Concurrent participation in other clinical study(ies) may be acceptable, with approval by the investigator and sponsor.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male and Females at least 14 years of age at the time of informed consent and sexually active.
Sampling Method: Probability Sample
Enrollment: 1912 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reid, PhD, Study Director — Gen-Probe, Incorporated
Locations (7):
- United States (7):
  - Wishard Health Services Department of Pathology Wishard Health Services, Indianapolis, Indiana
  - Louisiana State University Health Center, New Orleans, Louisiana
  - New England Center for Clinical Research, Fall River, Massachusetts
  - University of North Carolina Chapel Hill STD Clinic, Chapel Hill, North Carolina
  - Planned Parenthood Northeast Ohio, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center Division of Pediatric & Adolescent Gynecology, Cincinnati, Ohio
  - Planned Parenthood Houston and Southeast Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1912 male and female subjects were enrolled under this protocol. Of the 1912 subjects, 1862 were evaluable for analysis of CT or GC performance (conclusive infected status and at least one valid PANTHER Combo 2 Assay result)
Pre-assignment Details: Fifty (50) of the 1912 eligible subjects did not have a conclusive infected status or a valid Panther Combo 2 Assay result and are not included in the results below.
Groups:
- Positive Infected Status; Negative Infected Status: The Infected status algorithm used results from two specimen types and two reference types and two reference Nucleic Acid Amplification Tests (NAATs). Subjects were categorized as infected if a positive result occurred in each of the two reference NAATs. For female subjects, if positive NAAT result occurred only in the urine specimens and not in PreservCyt solution liquid pap specimens, the subject was categorized as infected; however for the evaluation of the non-urine specimen types, the specimens were considered non-infected. Subjects that could not be categorizes as infected or non-infected were excluded from the performance analyses.
Period: Overall Study
Arm/Group | Positive Infected Status | Negative Infected Status
Started | 264 | 1598
Completed | 264 | 1598
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Symptomatic and asymptomatic men (n=549) and women (n=1313) enrolled from seven geographically and ethnically diverse US clinical sites, including obstetrics and gynecology, family planning, public health, and STD clinics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Infected Status | Negative Infected Status | Total
Number analyzed (Participants) | 264 | 1598 | 1862
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 146 | 176
  Between 18 and 65 years | 234 | 1449 | 1683
  >=65 years | 0 | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (5.5) | 28.1 (9.8) | 27.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 1170 | 1313
  Male | 121 | 428 | 549
Region of Enrollment [Number; unit: participants]
  United States | 264 | 1598 | 1862

OUTCOME MEASURES:

1. Primary Outcome: APTIMA Combo 2 Assay Accuracy Compared to Infected Status by Sample Type
Description: Count of participants having a positive or negative APTIMA Combo 2 assay result (sensitivity and specificity)
Time Frame: Baseline
Population: Results for 4 gender-specific sample types were reported for 2 targets (CT, Chlamydia trachomatis; and GC, Neisseria gonorrhoeae infection). In this observational study, 1313 females (143 CT and/or GC-infected) and 549 males (121 CT and/or GC infected) contributed to one or more analyses.
Measure: Number; unit: participants
Arm/Group | Positive Infected Status | Negative Infected Status
Number analyzed (Participants) | 264 | 1598
participants
  Vaginal Swab for CT, AC2 pos (females) | 104 | 18
  Vaginal Swab for CT, AC2 neg (females) | 3 | 1149
  PreservCyt for CT, AC2 pos (females) | 112 | 0
  PreservCyt for CT, AC2 neg (females) | 2 | 1197
  Endocervical Swab for CT, AC2 pos (females) | 104 | 8
  Endocervical Swab for CT, AC2 neg (females) | 3 | 1139
  Urethral Swab for CT, AC2 pos (males) | 100 | 4
  Urethral Swab for CT, AC2 neg (males) | 0 | 445
  Vaginal Swab for GC, AC2 pos (females) | 42 | 5
  Vaginal Swab for GC, AC2 neg (females) | 1 | 1210
  PreservCyt for GC, AC2 pos (females) | 43 | 0
  PreservCyt for GC, AC2 neg (females) | 0 | 1250
  Endocervical Swab for GC, AC2 pos (females) | 42 | 2
  Endocervical Swab for GC, AC2 neg (females) | 0 | 1194
  Urethral Swab for GC, AC2 pos (males) | 34 | 0
  Urethral Swab for GC, AC2 neg (males) | 0 | 512

ADVERSE EVENTS:
Groups:
- Positive Infected Status; Negative Infected Status: The Infected status algorithm used results from two specimen types and two reference types and two reference Nucleic Acid Amplification Tests (NAATs). Subjects were categorized as infected if a positive result occurred in each of the two reference NAATs. For female subjects, if positive NAAT result occurred only in the urine specimens and not in PreservCyt solution liquid pap specimens, the subject was categorized as infected; however for the evaluation of the non-urine specimen types, the specimens were considered non-infected. Subjects that could not be categorized as infected or non-infected were excluded from the performance analyses
Arm/Group | Positive Infected Status | Negative Infected Status
Serious Adverse Events (participants affected / at risk) | 0/264 | 0/1598
Other Adverse Events (participants affected / at risk) | 0/264 | 0/1598

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less